CLINICAL TRIAL: NCT05726656
Title: Effect of Wii-console Based Exercise on Shoulder Range of Motion for Post-mastectomy
Brief Title: Effect of Wii-console Based Exercise on Shoulder Range of Motion for Post-mastectomy Lymphedema Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, doaa atef, lecturer of physical therapy for surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004199
Record Dates: First submitted 2023-02-03; First posted 2023-02-14 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Postmastectomy Lymphedema
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wii console based exercise group (Experimental): the patient will recieve wii console based exercise in addition to traditional physical therapy session
  Interventions: Other: traditional physical therapy session; Other: wii console based exercise
- control group (Other): the patient will recieve only the traditional physical therapy session
  Interventions: Other: traditional physical therapy session

INTERVENTIONS:
Other: traditional physical therapy session — manual lymph drainage-pneumatic compression and skin care
Other: wii console based exercise — execise session using the wii console video games
  Arms: wii console based exercise group

SUMMARY:
PURPOSE: To determine the effect of wii-console based exercise on shoulder ROM of both sides for post-mastectomy patients, and highlighting the effect of dominancy.

DETAILED DESCRIPTION:
Breast cancer has been the focused of many studies because it significantly affects both in developed and developing countries worldwide (Cameirão et al, 2008).

Lymphedema affects the range of motion of shoulder causing disability and affection of function.

Wii-console systems can be used as training tools to promote intensive training directed towards specific deficits and guide the patients in task-oriented activities. Moreover, it allows a real-time high-resolution monitoring, where is possible to have a quantitative assessment of relevant properties of the impairment, performance and recovery. On the other hand, virtual reality environment demand focus and attention of the patient, motivate the patient to perform the exercises, and provide a sense of achievement to the user (Torre et al, 2015).

HYPOTHESES:

The wii-console based exercise will have no effect on shoulder ROM for post-mastectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* All the patients will be females.
* Patients undergone mastectomy with lymph nodes dissection.
* all developed lymphedema after the surgery.

Exclusion Criteria:

* Vision problems.
* Medically instable patients.
* Balance disorders.
* Other musculoskeletal condition of shoulders.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
shoulder range of motion | 4 weeks
  flexion, extension, abduction, adduction , internal rotation and external rotation

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A Atef, PHD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No